CLINICAL TRIAL: NCT04148118
Title: A Phase 1 Randomized, Observer-Blind, Active- and Placebo-Controlled Dose Comparison, Safety, Tolerability and Immunogenicity Study of Intranasal Adjuvanted Anthrax Vaccine (BW-1010; rPA + 20%W805EC) in Healthy Adult Volunteers Administered by Nasal Sprayer and Pipette With an Additional Unblinded Positive Control Arm
Brief Title: A Safety and Immunogenicity of Intranasal Nanoemulsion Adjuvanted Recombinant Anthrax Vaccine in Healthy Adults
Acronym: IN NE-rPA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: BlueWillow Biologics (Industry)
Collaborators: Porton Biopharma Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: BW1010-001; HHSN272201600045C (Other Grant/Funding Number: NIAID); 16-0111 (Other: DMID Protocol Number)
Record Dates: First submitted 2019-10-28; First posted 2019-11-01 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Anthrax
Keywords: Anthrax; Nanoemulsion adjuvant; Nasal Vaccine; Recombinant Protective Antigen
MeSH Terms: conditions — Anthrax | interventions — Sodium Chloride; Biothrax

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to receive BW-1010 in 2 different dose levels (50 µg or 100 µg rPA), using 2 different method of administration (Aptar sprayer or pipette dropper). Negative control participants (Placebo) will receive saline using the 2 different methods as well. The positive control participants will receive BioThrax subcutaneously.
  Since this is first in humans, a sentinel group, 4 participants with the smaller dose level (50 µg rPA) and 2 placebos, will be dosed first. The main group of the 50 µg rPA and the higher level rPA sentinels will dosed after day 8 safety clearance of the low dose rPA sentinel participants.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The study participants and the study site personnel managing the participants will be blinded to the identity of the test article. The pharmacist and/or the pharmacy technician or non-study nurse at the study site will not be blinded and will be responsible for preparing, labeling, and administering the investigational product. During study drug administration, all the blinded personnel will be excluded from the vaccine administration site. In addition, participants will be asked to close their eyes or be offered the option of wearing a loose-fitting eye mask during the administration of the test article.
  Participants in the study arm that receive BioThrax SC and the clinical trial personnel that are managing them will not be blinded for this arm due to the different route of administration that makes blinding impossible. For laboratory and immunological testing, samples from participants receiving BioThrax will be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- NE+50µg rPA - sprayer (Experimental)
  Interventions: Biological: BW-1010: 50 µg - sprayer - IN
- NE+50µg rPA - pipette (Experimental)
  Interventions: Biological: BW-1010: 50 µg - pipette - IN
- NE+100µg rPA - sprayer (Experimental)
  Interventions: Biological: BW-1010: 100 µg - sprayer - IN
- NE+100µg rPA - pipette (Experimental)
  Interventions: Biological: BW-1010: 100 µg - pipette - IN
- Saline - sprayer (Placebo Comparator)
  Interventions: Biological: Saline (Placebo) - sprayer - IN
- Saline - pipette (Placebo Comparator)
  Interventions: Biological: Saline (Placebo) - pipette - IN
- BioThrax - SC (Active Comparator)
  Interventions: Biological: BioThrax (positive control) - SC

INTERVENTIONS:
Biological: BW-1010: 50 µg - sprayer - IN — 20% Nanoemulsion and 50 µg recombinant protective antigen administered intranasally by Aptar Bidose Sprayer (400µL).
  Two doses administered 4 weeks apart.
  Arms: NE+50µg rPA - sprayer
Biological: BW-1010: 50 µg - pipette - IN — 20% Nanoemulsion and 50 µg recombinant protective antigen administered intranasally by pipette (400µL).
  Two doses administered 4 weeks apart.
  Arms: NE+50µg rPA - pipette
Biological: BW-1010: 100 µg - sprayer - IN — 20% Nanoemulsion and 100 µg recombinant protective antigen administered intranasally by Aptar Bidose Sprayer (400µL)
  Two doses administered 4 weeks apart
  Arms: NE+100µg rPA - sprayer
Biological: BW-1010: 100 µg - pipette - IN — 20% Nanoemulsion and 100 µg recombinant protective antigen administered intranasally by pipette (400µL).
  Two doses administered 4 weeks apart.
  Arms: NE+100µg rPA - pipette
Biological: Saline (Placebo) - sprayer - IN — Saline (negative control) administered intranasally by Aptar Bidose Sprayer (400µL).
  Two doses administered 4 weeks apart.
  Arms: Saline - sprayer
Biological: Saline (Placebo) - pipette - IN — Saline (negative control) administered intranasally by pipette (400µL).
  Two doses administered 4 weeks apart.
  Arms: Saline - pipette
Biological: BioThrax (positive control) - SC — BioThrax licensed vaccine administered subcutaneously (500µL).
  Three doses administered 2 weeks apart.
  Arms: BioThrax - SC

SUMMARY:
The purpose of this clinical trial is to evaluate the safety and immunogenicity of BW-1010.

BW-1010 is a nanoemulsion adjuvanted recombinant protein (rPA) that would protect against fatal outcome resulting from exposure to anthrax.

The vaccine will be administered intranasally (IN) to healthy adults, age 18 - 49.

The study will be conducted in 84 volunteers in one center in the United States.

The study will compare 2 different dose levels of rPA (50µg and 100µg rPA), and 2 different administration methods (a sprayer and dropper) with a negative control (saline) and a positive control (the injectable BioThrax licensed vaccine).

The vaccines and negative controls will be administered in 2 IN doses (4 weeks apart). The positive control will be 3 subcutaneous doses, 2 weeks apart. All volunteers will be observed for 1 year after the last dose.

Immunological outcome studied will be from the serum, blood cells and nasal washes.

DETAILED DESCRIPTION:
This study is a single center, randomized, observer-blind, active- and placebo-controlled, dose comparison study to assess the safety, tolerability and immunogenicity of BW-1010 administered IN using an Aptar Bidose sprayer or an Eppendorf Electronic Repeater pipette in healthy adult volunteers. There is an additional unblinded BioThrax arm administered by SC injection. BioThrax is included in the study design only to provide a licensed, active control for immunogenicity and safety comparisons. A total of 84 participants will be enrolled in the study. Participants will be randomized in one of the following 7 arms:

A) BW-1010: 50µg - sprayer - IN, 400 µL; 16 participants.

B) BW-1010: 50µg - pipette - IN, 400 µL; 16 participants.

C) BW-1010: 100µg - sprayer - IN, 400 µL; 16 participants.

D) BW-1010: 100µg - pipette - IN, 400 µL; 16 participants.

E) Saline (Placebo) - sprayer - IN, 400 µL; 6 participants.

F) Saline (Placebo) - pipette - IN, 400 µL; 6 participants.

G) BioThrax (Positive control) - SC, 500 µL; 8 participants.

All participants receiving test article or placebo will receive two doses of the vaccine four weeks apart. Each of these participants will receive treatment intranasally using either an Aptar Bidose sprayer or an Eppendorf Electronic Repeater pipette. Eight participants will be randomized to receive a positive control (BioThrax vaccine) and will receive 3 doses of vaccine two weeks apart.

Since this is the first-in-human study for BW-1010, a total of twelve sentinel participants will receive either the test article or the placebo in a randomized fashion prior to dosing the main participants. Four of the 50 µg rPA vaccine and two placebo control participants will be randomized and dosed first, with no more than one participant/day with at least 24 hours safety follow up prior to enrolling the next participant. The Safety Review Committee (SRC) will review all safety data available through the Day 8 visit of the last sentinel participant dosed from this group and provide clearance to proceed with the 50 µg rPA Main Study participants and the 100 µg sentinel group. Four of the 100 µg rPA vaccine Sentinel Group and two placebo control participants will be randomized and dosed after safety clearance of the 50 µg rPA sentinel group, with no more than one participant/day with at least 24 hours safety follow up prior to enrolling the next participant. The SRC will review all safety data available through the Day 8 visit of the last sentinel participant dosed from this group and provide clearance to proceed with the 100 µg rPA Main Study participants.

Participants will be followed up for safety and tolerability for 1 year following last immunization.

Participants will be assessed for production of specific antibodies in the form of serum toxin neutralization antibodies (TNA) and serum anti-rPA IgG throughout the study until the termination visit.

Since this is a nasal vaccine and it is anticipated that the immune response will be different that the standard parental vaccines, the participants will be tested 10 days post last dose for rPA-specific cytokine on T-cells (IFN-ɤ, IL-5 and IL-17) and rPA-specific IgG and Ig-A on B-cells. Nasal wash will also be tested for total IgA and rPA-specific IgG and IgA.

Safety and immunogenicity analysis will include all randomized participants. Analysis will compare the different dose levels, different method of administration. Participants who received BW-1010 will be compared to participants who received the saline negative control and the BioThrax positive control.

COVID-19 Shut Down Impact on the Clinical Trial:

After the majority of the 50µg subjects had received only 1 of the 2 planned immunization, the Covid-19 pandemic stay-at-home order was instated and they could not receive their 2nd immunization. As a result of this, after COVID shut down was released, subjects involved in the clinical trial were divided into 2 Cohorts:

1. Cohort 1: Subjects from the Sentinel and 50µg main groups who received 2 or 1 immunizations prior to COVID-19 stay-at-home restrictions. Except for COVID-interrupted visits, these subjects will continue safety assessment at their their originally planned visits. Due to incomplete immunization schedule, no immunological testing will be performed.
2. Cohort 2: These are the subjects who were not enrolled prior to the Covid-19 impacts. In order to maintain enough power to detect critical safety issues in the clinical trial, these remaining 43 subjects will be randomized to receive the 100 µg rPA dose or placebo (either by pipette or sprayer) or BioThrax. No additional 50 µg rPA subjects will be dosed. These 43 subjects will follow the original study plan:

   1. Immunization at Week 0 and Week 4 (+ Week 2 for BioThrax).
   2. Follow up on Weeks 1, 5.5, 8, 12, 28 and 56 for safety and immunogenicity.

ELIGIBILITY:
Inclusion Criteria:

1. Between 18 to 49 years of age, inclusive.
2. Female of child-bearing potential, must be non-lactating and non-pregnant as confirmed by a negative serum pregnancy test conducted at screening and a negative urine pregnancy test conducted at the site within 24 hours preceding each receipt of vaccine.
3. Females should be either:

   1. Surgically sterile. Surgical sterilization includes hysterectomy, bilateral salpingectomy, tubal ligation or successful other permanent sterilization methods such as Essure® placement with documented confirmation test at least 3 months after the procedure, or
   2. At least one year post-menopausal, or
   3. Agree to use highly effective hormonal contraceptive method defined by a <1% failure rate that is not affected by adherence such as progestin releasing subdermal implants, or levonorgestrel releasing IUDs, for a minimum of 30 days prior to immunization and for 3 months following the last immunization. Concurrent use of a barrier method of birth control is not required. or
   4. If using a moderately effective contraceptive method defined by a 5-9% failure rate per year with typical use, such as the pill, hormone releasing transdermal patch or ring, or Progestin-only Injectable Contraceptive (DMPA) injections. Concurrent use of a barrier method of contraception is required. or
   5. Have acceptable sexual abstinence as defined by refraining from heterosexual intercourse for a minimum of 30 days prior to immunization and a credible intent to continue to do so until 3 months following the last immunization. The reliability of sexual abstinence will be to be evaluated in relation to the preferred and usual lifestyle of the subject.
4. Males must agree to use condoms from screening through 3 months following the last immunization, unless vasectomized.
5. Males must not donate sperm from screening through 3 months following the last immunization.
6. Are healthy, as determined by medical history, physical examination, vital signs, and clinical laboratory examinations. Healthy participants have no chronic medical conditions and no acute medical conditions that required the use of systemic prescription medications in the last 30 days or 5 half-lives, whichever is longer.
7. Comprehends the study requirements, is available for the required study period, and is able to attend scheduled visits.
8. Has given written informed consent to participate in the study.

Exclusion Criteria:

1. Presence of significant acute illness or any chronic medical condition.
2. Presence of psychiatric illness, currently untreated or clinically unstable (in the opinion of the PI) schizophrenia, bipolar disease, or other psychiatric diagnosis that may interfere with participant compliance or safety evaluations.
3. Participants with a history of chronic cough, reactive airway disease, asthma, chronic obstructive pulmonary disease (COPD), frequent sinus infections, sinusitis, allergic rhinitis, nasal polyps or obstruction, including deviated septum or other major nasopharyngeal anatomic abnormalities significant enough to obstruct the nasal openings, are to be excluded. Participants with seasonal rhinitis may be included if their 'season' does not occur within 3 months of the immunization date and they are not currently receiving intranasal steroids.
4. History of natural anthrax infection.
5. Receipt of any licensed or experimental anthrax vaccine at any time in the participant's lifetime.
6. The participant or an immediate household member is meeting criteria for which receipt of licensed anthrax vaccine is recommended or expected including:

   1. Exposure to animal products such as hides, hair, or bones which come from anthrax endemic areas and may be contaminated with Bacillus anthracis spores.
   2. Engagement in diagnostic or investigational activities which may result in contact with B. anthracis spores.
   3. Holding of a position such as veterinarians and others handling potentially infected animals.
   4. Military personnel for whom immunization with anthrax vaccine is required.
7. Positive serology for HIV-1 or HIV-2, or HCV antibodies.
8. Platelet count <150,000/mm3.
9. Fever >100.4°C within one week of immunization; this is considered as a temporary exclusion, as an otherwise eligible participant may be immunized once the fever has resolved. Participants must remain within the screening window or be rescreened if >30 days elapses prior to enrollment.
10. History of aspiration, dysphagia, swallowing disorders, stroke or other neurologic conditions that may predispose the participant to aspiration of test articles into the respiratory tract.
11. History of Bell's palsy.
12. Cancer or treatment for cancer, within 3 years. Participants with a history of cancer who are disease-free without treatment for 3 years or more are eligible. Participants with basal cell carcinoma or squamous cell carcinoma are allowed, unless present on or near the nose.
13. Impaired immune responsiveness, regardless of cause, including diabetes mellitus.
14. Known or suspected active chronic autoinflammatory condition
15. Presently receiving or a history of receiving any medications or treatments that affect the immune system such as immunoglobulin, interferon, immuno-modulators, cytotoxic drugs or drugs known to be frequently associated with significant major organ toxicity, or systemic corticosteroids (oral or injectable) in the past six (6) months.
16. Chronic use of inhaled or intranasal sprays including decongestants and corticosteroids; chronic use of these products is prohibited during the first 12 weeks of the study.
17. Presently a vaper, smoker or tobacco user or with a history of vaping, smoking or tobacco use within the past year prior to screening.
18. Receipt or planned administration of a non-study vaccine within 30 days of screening or 60 days after the initiation of the study. Immunization on an emergency basis such as with Tetanus Toxoids Adsorbed for adult use (Td or Tdap) upon exposure will be allowed. Administration of study vaccine can be delayed if a non-study vaccine has been administered and will be given as soon as acceptable, as described above.
19. Known allergy to any vaccine component.
20. History of allergic and/or anaphylactic type reaction to tetracycline-based drugs, injected vaccines, or to any of the components of BW-1010 [soybean oil, dehydrated alcohol (anhydrous ethanol), polysorbate 80 (Tween 80) and, Cetylpyridinium chloride (CPC)], or any of the BioThrax components (aluminium, benzethonium chloride, or formaldehyde).
21. History of drug or chemical abuse in the year before the study.
22. Receipt of any investigational product or nonregistered drug within the 30 days of screening, or currently enrolled in any investigational drug study, or intends to enroll in such a study within the ensuing 12 month period.
23. Use of nasally administered prescription or nasally administered over-the-counter (OTC) medications within seven (7) days before immunization.
24. Receipt of blood or blood products eight (8) weeks before study entry or planned receipt within the ensuing 12 month period.
25. Donation of blood or blood products within eight (8) weeks before screening or planned donation within the ensuing Week 12 visit.
26. Acute disease within a week prior to immunization, defined as the presence of a moderate or severe illness (as determined by the PI through medical history and physical examination) with or without fever. For participants with a minor illness, such as diarrhea, or mild upper respiratory tract infection with or without low-grade febrile illness, the participant can be re-screened once they have completely recovered.
27. Any condition that, in the opinion of the PI, might interfere with study objectives.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2020-01-08 (Actual); Primary Completion 2021-09-02 (Actual); Study Completion 2021-09-02 (Actual)

PRIMARY OUTCOMES:
Safety Objectives: Frequency of solicited systemic and local reactions (reactogenicity and tolerability) reported after each immunization | Up to Day 39 scheduled visit.
  This will be conducted throughout the 2 hours in-clinic observation following each immunization, during the follow up Safety Phone Call conducted 1-3 days post immunization, during the review of the Symptom Diary Reminder Card that will be distributed to participants following immunization and during the 7 to 10 day visit following each immunization.
Safety Objectives: Frequency of Adverse Events (AE) | Up to Day 85 scheduled visit.
  All treatment-emergent AEs will be summarized. These are AEs beginning or worsening after the initiation of the first immunization. These including any clinical laboratory abnormalities.
Safety Objectives: Frequency of Serious Adverse Events (SAEs) | Up to Day 393 scheduled visit.
  An adverse event is considered "serious" if it results in death, or a life-threatening AE, or in hospitalization, or in a substantial disruption of the ability to conduct normal life functions, or in a congenital anomaly/birth defect.
Primary Immunogenicity Objectives: Assess and compare the increase in rPA neutralizing antibodies following the different interventions in Cohort 2 subjects. | Day 57 and Day 85 (co-primary end point). The two time points will be compared to identify the optimum timing of peak immuneresponse following nasal vaccination.
  Use serum Toxin Neutralizing Assay (TNA) to compare immune response in the rPA 100 µg dose between the two different methods of administration (Aptar Bidose sprayer and Eppendorf Electronic Repeater pipette) of BW-1010 and compare them with the positive control arm receiving BioThrax.

SECONDARY OUTCOMES:
Secondary Immunogenicity Objectives: Assess and compare the increase in anti-rPA antibodies following the different interventions in Cohort 2 subjects. | Day 57 and Day 85.
  Use serum anti-rPA (ELISA) to compare immune response in the rPA 100 µg dose between two different methods of administration (Aptar Bidose sprayer and Eppendorf Electronic Repeater pipette) of BW-1010 and compare them with the positive control arm receiving BioThrax.

OTHER OUTCOMES:
Exploratory Immunogenicity Objectives: Assess and compare the increase in rPA neutralizing and anti-rPA antibodies following the different interventions in Cohort 2 subjects. | Baseline, Days 39, 197 and 393.
  Use serum TNA and anti-rPA (ELISA) to compare immune response in the 100 µg dose between two different methods of administration (Aptar Bidose sprayer and Eppendorf Electronic Repeater pipette) of BW-1010 and compare them with the positive control arm receiving BioThrax.
Exploratory Immunogenicity Objectives: Assess and compare the increase in mucosal antibodies following different interventions in Cohort 2 subjects. | Baseline and Day 39.
  Use nasal wash (NW) to assess mucosal antibody response (as measured by anti-rPA IgA, anti-rPA IgG and total mucosal IgA in NW) to compare mucosal immune response in the rPA 100 µg dose between the two different methods of administration (Aptar Bidose sprayer and Eppendorf Electronic Repeater pipette) of BW-1010 and compare them with the positive control arm receiving BioThrax.
Exploratory Immunogenicity Objectives: Assess and compare the increase in cell meditated immune responses in PBMCs following different interventions in Cohort 2 subjects. | Baseline and Day 39.
  Use PBMCs to assess cell-mediated immunity (CMI) (as measured by T-cell ELISpot for rPA-specific IL-17, IFN-γ and IL-5 and B-cell ELISpot for rPA-specific IgG and IgA) to compare CMI responses in the rPA 100 µg dose between two different methods of administration (Aptar Bidose sprayer and Eppendorf Electronic Repeater pipette) of BW-1010 and compare them with the positive control arm receiving BioThrax.

CONTACTS AND LOCATIONS:
Locations (1):
- Johnson County Clin-Trial, Lenexa, Kansas, United States

IPD SHARING:
Plan to Share IPD: No